CLINICAL TRIAL: NCT05150782
Title: The Effect of a Mixture of Micellized Curcumin/Boswellia Serrata/Ascorbic Acid on Health-related Quality of Life in Patients With Post-acute COVID-19 Syndrome.
Brief Title: The Effect of Micellized Food Supplements on Health-related Quality of Life in Patients With Post-acute COVID-19 Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PhysioMetrics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MyCellVSLongCOVID
Record Dates: First submitted 2021-12-05; First posted 2021-12-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Post-acute COVID-19 Syndrome
Keywords: micelles; dietary supplements
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Single-arm intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curcumin/Boswellia Serrata/Ascorbic acid mixture (Experimental): The daily intake of 2x10 drops of a mixture of micellized curcumin(2%), boswellia serrata (1,5%) and ascorbic acid (6%).
  Interventions: Dietary Supplement: Curcumin/Boswellia Serrata/Ascorbic acid mixture

INTERVENTIONS:
Dietary Supplement: Curcumin/Boswellia Serrata/Ascorbic acid mixture — The daily intake of 2x10 drops of a mixture of micellized curcumin (2%), boswellia serrata (1.5%) and ascorbic acid (6%).

SUMMARY:
Food supplements like curcumin and boswellia serrata have been used traditionally for anti-inflammatory purposes. A well-known problem of these substances in their natural form is the low bioavailability. Micellization of these substances has been shown to increase the bioavailability significantly and thereby the clinical efficacy. The clinical value of these micellized substances has been presented in numerous clinical studies and in particular in patients with acute COVID-19. This study aims to examine the effect of a mixture of micellized curcumin, boswellia serrata and ascorbic acid on patients with long COVID.

DETAILED DESCRIPTION:
The participants will be asked to take the micellized supplements daily, at home for 6 weeks. During this 6 weeks several questionnaires will be taken to asses general health-related quality of life. Follow-up measurements will be done at 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed SARS-CoV-2 infection at least 28 days prior to study participation
* Patients who are experiencing symptoms of PACS (with a PCFS of 1 or higher)
* 18 years or older and younger than 85
* Good understanding of written German

Exclusion Criteria:

* Currently under pharmacological treatment for PACS
* Any planned medical surgery or intervention where medication intake is necessary in the coming 14 weeks
* Allergy to curcumin or Boswellia
* Active malignancy
* Medical history of Human Immunodeficiency Virus (HIV) infection, or any serious immunocompromised state.
* Pregnancy (or planned pregnancy in the coming 14 weeks) ( - Patients who are taking anticoagulants or have diabetes type I or II are only allowed to participate if their general practitioner is informed)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-17 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life | Week 1, 2, 3, 4, 5, 6, 10 and 14.
  Health-related quality of life is measured with the 'Short-Form 12' (SF-12) from 0 to 100, where higher scores on the SF-12 represent better health-related quality of life.

SECONDARY OUTCOMES:
Change in patient selected functional limitations in daily life, measured with the 'Patient specific functional scale (PSFS). | Week 1, 2, 3, 4, 5, 6, 10 and 14.
  Patient specific limitations in daily life are measured with the 'Patient Specific Functional Scale' (PSFS). The scale is a visual analogue scale ranging from 0 to 100, with 0 meaning no limitations in the patient selected functional activity and 100 means it is impossible to perform this activity.
Change in general health status | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 , 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21
  Change in general health status is measured with a dichotomous yes or no question.
Change in general health | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 , 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21
  Percentage of change of general health is asked for, where 0 represents no change and 100% means complete change,
Change in Post COVID functional status measured with the 'Post COVID Functional Status' (PCFS). | Week 1, 2, 3, 4, 5, 6, 10 and 14.
  Self-Test for ordinal scaling of degree of post-COVID symptoms with 0 representing no symptoms and 4 several functional limitations.

OTHER OUTCOMES:
Course of general health | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 , 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21
  Graphical depiction of course of self-perceived change of general health.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Kangeldi, MSc, Study Director — Cognitive Health Platform AG

IPD SHARING:
Plan to Share IPD: Yes
Data are available for researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available as soon as the results are published. The availability of the data is 5 years.
Access Criteria: i) Affiliated researcher, 2) researcher must be able to demonstrate that accessing the raw study data is necessary to be able to conduct his/her research project